CLINICAL TRIAL: NCT01733381
Title: An Examination of the Differential Effects of Running Minimally Shod vs. in Shoes on Physiology and Emotional States Relevant to Major Depression.
Brief Title: Effects of Barefoot Running vs. in Shoes on Physiology and Mood
Status: Completed | Type: Observational
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Other Study IDs: 12-0370-02
Record Dates: First submitted 2012-11-14; First posted 2012-11-27 (Estimated); Last update posted 2025-07-31 (Actual); Status verified 2014-02

CONDITIONS: Autonomic Nervous System (ANS) Functioning and Mood State
Keywords: Barefoot running, minimally shod running, non-invasive measures of autonomic nervous system (ANS) functioning and mood state.

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Barefoot runners: This group of individuals will run in minimally shod foot ware. For the purposes of this study we have defined this to be Vibram Five Finger shoes. Participants will be runners who consistently run in these shoes at least 20 miles per week.
- Shoed runners: This group of individuals will run in normal running shoes. Participants will be runners who consistently run in regular running shoes (that are not considered by industry standards to be minimal shoes) at least 20 miles per week.

SUMMARY:
Aerobic exercise impacts bodily processes implicated in the pathophysiology of major depression. Consistent with these effects, aerobic exercise in general, and running in particular, has been repeatedly shown to have both immediate mood elevating and longer-term antidepressant effects. To the investigators' knowledge, all studies of running as a therapeutic intervention for mood have had subjects run in standard running shoes, despite increasing evidence that running barefoot or in shoes with minimal effect on foot strike (i.e. "minimally shod") leads to marked changes in how people run in ways that might have physiological effects of relevance to health. Thus, nothing is currently known about differences in effects on depression-relevant physiological or emotional functioning between running either barefoot or minimally-shod vs. running in standard running shoes (hereafter called "shoed). The current pilot study is designed to begin addressing these issues by examining effects of minimally shod vs. shoed running on non-invasive measures of autonomic nervous system (ANS) functioning and mood state.

DETAILED DESCRIPTION:
Aerobic exercise impacts bodily processes implicated in the pathophysiology of major depression. Consistent with these effects, aerobic exercise in general, and running in particular, has been repeatedly shown to have both immediate mood elevating and longer-term antidepressant effects. To the investigators' knowledge, all studies of running as a therapeutic intervention for mood have had subjects run in standard running shoes, despite increasing evidence that running barefoot or in shoes with minimal effect on foot strike (i.e. "minimally shod") leads to marked changes in how people run in ways that might have physiological effects of relevance to health. Thus, nothing is currently known about differences in effects on depression-relevant physiological or emotional functioning between running either barefoot or minimally-shod vs. running in standard running shoes (hereafter called "shoed). The current pilot study is designed to begin addressing these issues by examining effects of minimally shod vs. shoed running on non-invasive measures of autonomic nervous system (ANS) functioning and mood state. The investigators have selected the ANS as the physiological focus of the current study for several reasons including: 1) running acutely alters ANS activity; 2) running (and aerobic fitness in general) is associated with increased parasympathetic and reduced sympathetic activity at rest; 3) increased parasympathetic tone in the body has been repeatedly associated with emotional well-being and stress resilience, whereas reduced parasympathetic tone has been reliably associated with major depression; 4) given increasing evidence that ancestral humans may have run exceptionally long distances to hunt prey to exhaustion, it is likely that such running was conducted under fairly significant parasympathetic tone to reduce energy expenditure; 5) ancestral humans ran barefoot or minimally shod suggesting that the type of foot strike pattern encouraged by these styles of running may have enhanced parasympathetic tone compared to running with heel strike such as occurs when running shoed; and 6) therefore minimally shod running might differentially impact parasympathetic tone in ways that would make it more effective as a treatment for depression than running shoed.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female subjects between the ages of 18 and 45 at study entry (per a self report- females must be in the follicular phase of their menstrual cycle, within ~14 days of the end of their last period)
* Fully ambulatory and in good medical health (see exclusion criteria below for specifics)
* Ability to read/understand English
* Consistent practice of running at least three times a week for a total of at least 30 minutes at a time.

Exclusion Criteria:

* Potential subjects will be excluded for a diagnosis of any serious ongoing medical or psychiatric condition that might unduly influence results or increase risk of study participation, including but not limited to:

  * Malignancy
  * Auto-immune disorder
  * Cardiovascular disease (except treated hypertension)
  * Neurologic disorder
  * Endocrinopathy (other than treated hypothyroidism)
  * Chronic infection (i.e. human immunodeficiency virus, hepatitis B or C)
  * Any renal, hepatic or hematological abnormality (other than history of mild anemia)
  * Current major depression or major depression requiring hospitalization or resulting in suicide attempt in past year.
* Subjects will also be excluded for use of medications that might impact ANS functioning, including but not limited to beta-blockers, calcium channel blockers and alpha-blockers, and any medication with anticholinergic properties (e.g., many antihistamines).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Avid barefoot runners and regular 'shoed' runners will be selected from local running groups and clubs.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2012-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
To examine whether running minimally-shod produces changes in ANS function both during and after running when compared to running shoed. | Day 1 (Running day - no change is being assessed, participants run only ONCE during the study)
  Hypothesis 1: For any given amount of energy expenditure, running minimally shod will be associated with increased indices of parasympathetic tone when compared to running in shoes.
  Hypothesis 2: In all subjects, for any given amount of energy expenditure, the degree of forwardness of foot strike (i.e. toward toes and away from heel) will be correlated with increased measures of parasympathetic tone during and following running.

SECONDARY OUTCOMES:
Specific Aim 2: To examine whether running minimally-shod produces changes in emotional state both during and after running when compared to running shoed. | Day 1 (Running day - no change is being assessed, participants run only ONCE during the study)
  Hypothesis 3: For any given amount of energy expenditure, running minimally shod will be associated with increased self-reported positive mood and reduced negative mood when compared to running in shoes.
  Hypothesis 4: In all subjects, for any given amount of energy expenditure, the degree of forwardness of foot strike (i.e. toward toes and away from heel) will be correlated with increased self-reported positive mood and reduced negative mood.
To examine whether changes in ANS activity associated with running are associated with changes in mood. | Day 1 (Running day - no change is being assessed, participants run only ONCE during the study)
  Hypothesis 5: Parasympathetic tone both during and following running will be associated with self-reported mood both during and following running.

CONTACTS AND LOCATIONS:
Locations (1):
- Human Evolutionary Biomechanics Laboratory in the Park Student Union, Room 236 at the University of Arizona, Tucson, Arizona, United States